CLINICAL TRIAL: NCT01142713
Title: The Impact of Patient Positioning and Use of Belly Board on Small Bowel and Urinary Bladder Volume Irradiated in Patients Receiving Radiotherapy for Rectal Cancer: A Prospective Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Eliahu Gez MD, TASMC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-EG-0681-09-TLV-CTIL
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-02

CONDITIONS: Rectal Cancer
Keywords: Small Bowel Radiotherapy Dose; This is a prospective non-randomized open study to evaluate the impact of patient's positioning and use of belly board in rectal radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

INTERVENTIONS:
Radiation: Patient Position During Radiotherapy — Two simulations, one in the supine position on a flat table and another in the prone position on belly board

SUMMARY:
Radiotherapy has a significant impact on local control, disease free survival and overall survival in patients with rectal cancer T2, N1, M0 and T3-4, any N, M0. Treatment is accompanied by side effects, mainly due to the inclusion of the small bowel and urinary bladder in the treatment fields.

Two major modalities have been pursued to reduce the volume of small intestine and urinary bladder in treatment volume. One is a surgical procedure, such as absorbable mesh. These procedures have failed implementation in daily clinical practice. The second modality aims to save the small intestine and urinary bladder from the toxicity of radiotherapy by modulating the radiotherapy planning procedure. Using the belly board and changing the standard position from supine to prone could achieve this aim; in part due to gravitational displacement of the bowel. Several studies have evaluated the impact of positioning and use of belly board in patients receiving pelvis irradiation for rectal cancer. The results are inconclusive, but the prone position with belly board appears promising.

This study carefully evaluates the impact of patient's positioning and belly board on dose volume histogram of small bowel and urinary bladder

DETAILED DESCRIPTION:
This is a prospective non-randomized open study to evaluate the impact of patient's positioning and use of belly board in rectal radiotherapy.

In contrast to previous studies, the clinical target volume and organ at risk will be contouring for three-dimensional planning. With the aid of modern imaging, correlation can be obtained between dose and volume (DVH) since both parameters have an impact on organ tolerance to ionizing radiation.

Thirty patients with rectal cancer scheduled to receive "rectal radiotherapy", pre or postoperative will be included (15 patients from each group).

In addition to radiotherapy, the patients will receive concomitant chemotherapy.

Chemotherapy: The chemotherapy will consist of one of the following:

1. Capecitabine (Xeloda) 825mg/m2 ×2/day, given every day of radiotherapy.
2. 5FU continuous infusion 180 mg/m2, D1-5/week X 5

Radiotherapy:

The clinical target volume (CTV) for preoperative radiotherapy will include the entire rectum and regional lymph nodes. The following lymph nodes will be contoured: peri rectal, pre sacral, obturator, internal iliac and distal common iliac. The contouring of the rectum will start 1 cm above the anal verge until the sigmoid (average 15 cm).

The planning target volume will be included in the CTV + 5mm The following organs at risk will be contoured: small intestine, urinary bladder and femoral joints.

The prescription dose will be: 180cGy/day, 5 times a week for a total 5,040cGy (38b fraction over 6 weeks.

Each patient will undergo two simulations, one in the supine position on a flat table and another in the prone position on belly board. No contrast media will be used. The urinary bladder will be full in an attempt to push the small bowel away from the treatment volume. Three dimensional conformal radiotherapy planning will be done twice (one in each position). Three and four fields plan will be evaluate in each position. Therefore a comparison will be between four plains and the optimal plan will be chose for treatment..

The following parameters will be calculated:

1. Total volume of the small bowel
2. Total volume of urinary bladder
3. Intersection of PTV Volume and of small bowel volume
4. Intersection of PTV volume and of urinary bladder volume
5. Volume of small bowel included in the treatment volume
6. Volume of urinary bladder in the treatment volume

ELIGIBILITY:
Inclusion Criteria:

* patients with rectal cancer scheduled to receive "rectal radiotherapy", pre or postoperative

Exclusion Criteria:

* No exclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Dose and irradiated volume of small bowel and urinary bladder | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Eliahu Gez, MD, Principal Investigator — TASMC; Elaihu Gez, MD, Study Chair — TASMC; Eliahu Gez, MD, Study Chair — TASMC
Locations (1):
- TASMC, Tel Aviv, Israel